CLINICAL TRIAL: NCT01032330
Title: A Randomized Clinical Trial of Observation Versus Occlusion Therapy for Intermittent Exotropia
Brief Title: Observation Versus Occlusion Therapy for Intermittent Exotropia
Acronym: IXT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: Pediatric Eye Disease Investigator Group (Network); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NEI-146; 2U10EY011751 (NIH)
Record Dates: First submitted 2009-12-11; First posted 2009-12-15 (Estimated); Results first posted 2019-05-08 (Actual); Last update posted 2020-05-19 (Actual); Status verified 2020-05

CONDITIONS: Exotropia
Keywords: intermittent exotropia; IXT; natural history; occlusion therapy; occlusion; patching; strabismus; strabismus treatment; stereoacuity; motor alignment
MeSH Terms: conditions — Exotropia; Bites and Stings; Strabismus

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Observation (No Intervention): Patients randomized to the observation group will receive no treatment (other than refractive correction).
- Occlusion Therapy (Active Comparator): Patients randomized to the occlusion treatment group will receive occlusion (patching) for 3 hours per day for at least 3 months. Choice of which eye to occlude, or whether to alternate daily, is at investigator's discretion.
  Interventions: Device: occlusion treatment

INTERVENTIONS:
Device: occlusion treatment — Patients randomized to the occlusion treatment group will receive occlusion (patching) for 3 hours per day for at least 3 months. Choice of which eye to occlude, or whether to alternate daily, is at investigator's discretion.
  Other Names: occlusion therapy; patching
  Arms: Occlusion Therapy

SUMMARY:
The present study is being conducted to assess the natural history of intermittent exotropia and to establish the effectiveness of occlusion in its treatment.

Study Objectives:

* To determine the effectiveness of occlusion for the treatment of intermittent exotropia among patients aged 3 to < 11 years who have baseline near stereoacuity of 400 arcsec or better by Preschool Randot stereotest
* To determine the natural history of intermittent exotropia among patients aged 3 to < 11 years who have baseline near stereoacuity of 400 arcsec or better by Preschool Randot stereotest

DETAILED DESCRIPTION:
Intermittent exotropia (IXT) is the most common form of childhood-onset exotropia with an incidence of 32.1 per 100,000 in children under 19 years of age. Intermittent exotropia is characterized by an exotropia that is not constant and is mainly present in the distance but may also be present at near. Many cases of IXT are treated using non-surgical interventions, such as part-time occlusion, fusional vergence exercises, and over-minus lenses. The rationale for such interventions is that they may improve the ability to control the IXT and preserve stereoacuity, thereby potentially addressing both visual function and social concerns, and may delay or eliminate the need for surgical correction of IXT. Nevertheless, the natural history of IXT is unknown and in many cases it is not known whether withholding treatment may in fact allow for spontaneous resolution or improvement in IXT, making non-surgical or surgical intervention unnecessary. Moreover, although non-surgical treatments for IXT are commonly prescribed, such treatments have not been subjected to rigorous study and their efficacy in improving visual function or social concerns remains unclear.

One aim of the present study is to better understand the natural history of IXT. Available reports on the natural history of IXT disagree on the progression of the disease. A 1966 study by von Noorden (cited in von Noorden and Campos) found that over an average of 3.5 years of follow-up, 75% of 51 patients showed signs of IXT progression, 9% showed no change, and 16% improved without therapy. A 1968 retrospective study by Hiles et al found that after a minimum of 6 years follow up with observation and nonsurgical treatment, 81% of 48 patients showed no change in angle of deviation. The results of more recent retrospective studies show some reporting that the majority of cases improve over time, others reporting that most cases remain stable, and still others reporting that most cases deteriorate. It is therefore unclear what proportion of patients, if left untreated, is likely to deteriorate, improve, or remain stable over time. Natural history data acquired during this study will help determine not only what proportion of patients change over time, but whether there are associated prognostic indicators of deterioration or improvement. Such data will not only enable better identification of those patients with IXT likely to benefit from treatment and those for whom treatment is likely to be unnecessary, but will also improve the quality of medical advice to parents regarding the likely progression of the disease, thus alleviating anxiety.

The aim of most forms of non-surgical treatments for IXT is to improve the strength and/or quality of binocular single vision by either eliminating suppression, increasing awareness of diplopia, and/or increasing positive fusional amplitudes. Commonly used non-surgical treatment methods include: occlusion, fusional vergence exercises (sometimes known as vision therapy or orthoptics), and over-minus lenses. When surveyed in 1990, members of the American Association for Pediatric Ophthalmology and Strabismus reported that occlusion was the most commonly used form of non-surgical treatment. More recently (2008), a poll of our investigator group revealed again that occlusion was the most widely prescribed non-surgical treatment for children affected by IXT.

Occlusion is thought to work by interrupting the development of or eliminating already present suppression, an adaptation to avoid diplopia in IXT. Persistent or entrenched suppression prevents normal binocular vision and may lead to permanent loss of stereoacuity. If successful, occlusion may then result in improved binocular sensory fusion.

As reported in recent reviews of treatment for IXT, previous studies of occlusion vary regarding the recommended occlusion dose (from 3 hours a day to full time), the optimum duration of occlusion treatment (from 6 weeks to 42 months), and which eye should be occluded (preferred/dominant eye or alternate eyes). For the majority of studies, part-time occlusion, rather than full-time occlusion was preferred. In the three occlusion studies conducted prospectively, the recommended dose was either 3 hours a day, 3 to 6 hours a day, or 4 to 6 hours a day, and the duration of occlusion ranged from 3 months to 6 months to up to 42 (mean 15) months. Nevertheless, these previous studies of occlusion for the treatment of IXT used a variety of outcome measures at a variety of non-standardized time points; therefore, no definite conclusions can be drawn from the existing literature.

Although occlusion treatment for IXT treatment is widely used, there have been no randomized clinical trials evaluating its effectiveness. Understanding the degree of effectiveness of occlusion treatment for IXT and the natural history of IXT has important public health implications. Successful restoration of binocular alignment and normal binocular function with occlusion therapy, or spontaneous improvement, will reduce the proportion of children undergoing surgery. Defining the rate of success with either occlusion or observation is therefore important in planning treatment for children with IXT. Alternatively, evidence of low treatment effectiveness with occlusion will help avoid unnecessary treatment.

The present study is being conducted to assess the natural history of IXT and to establish the effectiveness of occlusion in its treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 12 months to < 11 years
* Intermittent exotropia (manifest deviation) meeting all of the following criteria:

  * Intermittent exotropia at distance OR constant exotropia at distance and either intermittent exotropia or exophoria at near
  * Exodeviation at least 15PD at distance OR near measured by prism and alternate cover test (PACT)
  * Exodeviation at least 10PD at distance measured by PACT
* No previous surgical or non-surgical treatment for IXT (other than refractive correction)
* Visual acuity in the worse eye at least 0.3 logMAR (20/40 on ATS HOTV or 70 letters on E-ETDRS) for children ≥ 3 years of age
* No interocular difference of visual acuity more than 0.2 logMAR (2 lines on ATS HOTV or 10 letters on E-ETDRS) for children ≥ 3 years of age
* No hyperopia greater than +3.50 D spherical equivalent in either eye
* No myopia greater than -6.00 D spherical equivalent in either eye
* No prior strabismus, intraocular, or refractive surgery
* No abnormality of the cornea, lens, or central retina
* Investigator willing to observe the IXT untreated for 3 years unless specific criteria for deterioration are met

Exclusion Criteria:

* Pure phoria at both distance and near
* Prior non-surgical treatment for IXT other than refractive correction (e.g., vergence therapy, occlusion, vision therapy/orthoptics, or deliberate over-minus with spectacles more than 0.50D)
* Previous amblyopia treatment other than refractive correction within 1 year
* Vision therapy/orthoptics for any reason within the last year
* Interocular visual acuity difference more than 0.2 logMAR (2 lines on ATS HOTV for patients 3 to < 7 years old or 10 letters on E-ETDRS for patients ≥ 7 years old) (patients ≥ 3 years only) and/or investigator plans to initiate amblyopia treatment at this time.
* Limitation of ocular rotations due to restrictive or paretic strabismus
* Craniofacial malformations affecting the orbits
* Ocular disorders which would reduce visual acuity (except refractive error)
* Prior strabismus surgery or botulinum injection, intraocular surgery, or refractive surgery
* Strabismus surgery planned
* Known skin reactions to patch or bandage adhesives
* Significant neurological impairment such as cerebral palsy. Patients with mild speech delays or common reading and/or learning disabilities are not excluded.
* Investigator planning to change refractive correction at this time (if the patient is otherwise eligible, the investigator should consider prescribing refractive correction and bringing the patient back at a later time for enrollment)

Ages: 12 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 611 (Actual)
Dates: Start 2010-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan A Cotter, O.D., M.S., Study Chair — Southern California College of Optometry, Fullerton, CA; Brian G Mohney, M.D., Study Chair — Department of Ophthalmology, Mayo Clinic, Rochester, MN
Locations (2):
- United States (2):
  - Southern California College of Optometry, Fullerton, California
  - Mayo Clinic Department of Ophthalmology, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH data sharing policy, a de-identified database is placed in the public domain on the PEDIG public website after the completion of each protocol and publication of the primary manuscript.
Time Frame: The data from the 6-month study is entered. The data for the 3-year study will be made available in 2020.
Access Criteria: Users will need a valid email address
URL: https://public.jaeb.org/pedig/stdy/153

REFERENCES:
- [Result] Pediatric Eye Disease Investigator Group; Cotter SA, Mohney BG, Chandler DL, Holmes JM, Repka MX, Melia M, Wallace DK, Beck RW, Birch EE, Kraker RT, Tamkins SM, Miller AM, Sala NA, Glaser SR. A randomized trial comparing part-time patching with observation for children 3 to 10 years of age with intermittent exotropia. Ophthalmology. 2014 Dec;121(12):2299-310. doi: 10.1016/j.ophtha.2014.07.021. Epub 2014 Sep 16. PMID 25234012
- [Result] Pediatric Eye Disease Investigator Group; Mohney BG, Cotter SA, Chandler DL, Holmes JM, Chen AM, Melia M, Donahue SP, Wallace DK, Kraker RT, Christian ML, Suh DW. A Randomized Trial Comparing Part-time Patching with Observation for Intermittent Exotropia in Children 12 to 35 Months of Age. Ophthalmology. 2015 Aug;122(8):1718-25. doi: 10.1016/j.ophtha.2015.04.025. Epub 2015 Jun 11. PMID 26072346
- [Result] Pediatric Eye Disease Investigator Group; Writing Committee; Mohney BG, Cotter SA, Chandler DL, Holmes JM, Wallace DK, Yamada T, Petersen DB, Kraker RT, Morse CL, Melia BM, Wu R. Three-Year Observation of Children 3 to 10 Years of Age with Untreated Intermittent Exotropia. Ophthalmology. 2019 Sep;126(9):1249-1260. doi: 10.1016/j.ophtha.2019.01.015. Epub 2019 Jan 26. PMID 30690128
- [Result] Cotter SA, Mohney BG, Chandler DL, Holmes JM, Wallace DK, Melia BM, Wu R, Kraker RT, Superstein R, Crouch ER, Paysse EA; Pediatric Eye Disease Investigator Group. Three-year observation of children 12 to 35 months old with untreated intermittent exotropia. Ophthalmic Physiol Opt. 2020 Mar;40(2):202-215. doi: 10.1111/opo.12668. PMID 32202318
- [Derived] Pang Y, Gnanaraj L, Gayleard J, Han G, Hatt SR. Interventions for intermittent exotropia. Cochrane Database Syst Rev. 2021 Sep 13;9(9):CD003737. doi: 10.1002/14651858.CD003737.pub4. PMID 34516656
- [Derived] Holmes JM, Hercinovic A, Melia BM, Leske DA, Hatt SR, Chandler DL, Dean TW, Kraker RT, Enyedi LB, Wallace DK, Mohney BG, Cotter SA; Pediatric Eye Disease Investigator Group. Health-related quality of life in children with untreated intermittent exotropia and their parents. J AAPOS. 2021 Apr;25(2):80.e1-80.e4. doi: 10.1016/j.jaapos.2020.10.011. Epub 2021 Mar 8. PMID 33705917
- See also: PubMed Abstract - Older Cohort — https://www.ncbi.nlm.nih.gov/pubmed/25234012
- See also: PubMed Central HHS Public Access - Full Text - Older Cohort — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC4253733/
- See also: PubMed Abstract - Younger Cohort — https://www.ncbi.nlm.nih.gov/pubmed/26072346

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Aside from the two primary cohorts (older and younger), there were 52 patients in a separate exploratory cohort of patients who had little or no stereoacuity (800 or Nil); this cohort is not being reported based on the criteria listed in the protocol.
Groups:
- Older Cohort Observation Group: Older Cohort patients aged 3 to <12 years randomized to the observation group will receive no treatment (other than refractive correction).
- Older Cohort Occlusion Therapy Group: Occlusion treatment: Older cohort patients aged 3 to <12 years randomized to the occlusion treatment group will receive occlusion (patching) for 3 hours per day for at least 3 months. Choice of which eye to occlude, or whether to alternate daily, is at investigator's discretion.
- Younger Cohort Observation Group: Younger cohort patients aged 12 to 35 months randomized to the observation group will receive no treatment (other than refractive correction).
- Younger Cohort Occlusion Therapy Group: Occlusion treatment: Younger cohort patients aged 12 to 35 months randomized to the occlusion treatment group will receive occlusion (patching) for 3 hours per day for at least 3 months. Choice of which eye to occlude, or whether to alternate daily, is at investigator's discretion.
Period: Overall Study
Arm/Group | Older Cohort Observation Group | Older Cohort Occlusion Therapy Group | Younger Cohort Observation Group | Younger Cohort Occlusion Therapy Group
Started | 183 | 175 | 97 | 104
Completed | 165 | 151 | 87 | 90
Not Completed | 18 | 24 | 10 | 14

BASELINE CHARACTERISTICS:
Groups:
- Older Cohort Observation Group; Younger Cohort Observation Group: Patients randomized to the observation group will receive no treatment (other than refractive correction).
- Older Cohort Occlusion Therapy Group; Younger Cohort Occlusion Therapy Group: Occlusion treatment: Patients randomized to the occlusion treatment group will receive occlusion (patching) for 3 hours per day for at least 3 months. Choice of which eye to occlude, or whether to alternate daily, is at investigator's discretion.
- Total: Total of all reporting groups
Arm/Group | Older Cohort Observation Group | Older Cohort Occlusion Therapy Group | Younger Cohort Observation Group | Younger Cohort Occlusion Therapy Group | Total
Number analyzed (Participants) | 183 | 175 | 97 | 104 | 559
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 183 | 175 | 97 | 104 | 559
  Between 18 and 65 years | 0 | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 6.1 (2.0) | 5.9 (2.0) | 2.0 (0.54) | 2.0 (0.57) | 6.0 (2.0)
Age, Customized [Count of Participants; unit: Participants]
  3 to <5 years | 61 | 68 | 0 | 0 | 129
  5 to <7 years | 67 | 64 | 0 | 0 | 131
  7 to <9 years | 33 | 26 | 0 | 0 | 59
  9 to <11 years | 22 | 17 | 0 | 0 | 39
  1 to <1.5 years | 0 | 0 | 22 | 23 | 45
  1.5 to <2 years | 0 | 0 | 28 | 18 | 46
  2 to <2.5 years | 0 | 0 | 24 | 34 | 58
  2.5 to <3 years | 0 | 0 | 23 | 28 | 51
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 98 | 58 | 66 | 337
  Male | 68 | 77 | 39 | 38 | 222
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 112 | 109 | 65 | 60 | 346
  Black/African American | 23 | 25 | 13 | 14 | 75
  Hispanic or Latino | 32 | 22 | 13 | 21 | 88
  Other | 14 | 13 | 6 | 9 | 42
  Unknown/not reported | 2 | 6 | 0 | 0 | 8
Average Visual Acuity [Count of Participants; unit: Participants] — This measure was used exclusively with the older cohort, no data reported on this characteristic for the younger cohort.
  Participants
    20/12 or 20/16 | 21 | 22 | 0 | 0 | 43
    20/20 | 65 | 70 | 0 | 0 | 135
    20/25 | 73 | 45 | 0 | 0 | 118
    20/32 | 17 | 28 | 0 | 0 | 45
    20/40 or worse | 7 | 6 | 0 | 0 | 13
Average Visual Acuity [Mean (Standard Deviation); unit: logMAR] — Population: This measure was used exclusively with the older cohort, no data reported on this characteristic for the younger cohort.
  logMAR
    number analyzed (Participants) | 183 | 175 | 0 | 0 | 358
    (all) | 0.04 (.09) | 0.04 (.10) |  |  | 0.04 (0.10)
Interocular difference in visual acuity (lines) [Count of Participants; unit: Participants] — Population: This measure was used exclusively with the older cohort, no data reported on this characteristic for the younger cohort.
  Participants
    0: number analyzed (Participants) | 183 | 175 | 0 | 0 | 358
    0 | 86 | 85 |  |  | 171
    >0 to<1: number analyzed (Participants) | 183 | 175 | 0 | 0 | 358
    >0 to<1 | 45 | 37 |  |  | 82
    1: number analyzed (Participants) | 183 | 175 | 0 | 0 | 358
    1 | 42 | 43 |  |  | 85
    >1 to<2: number analyzed (Participants) | 183 | 175 | 0 | 0 | 358
    >1 to<2 | 4 | 5 |  |  | 9
    2: number analyzed (Participants) | 183 | 175 | 0 | 0 | 358
    2 | 6 | 1 |  |  | 7
Interocular difference in visual acuity (lines) [Mean (Standard Deviation); unit: logMAR] — Population: This measure was used exclusively with the older cohort, no data reported on this characteristic for the younger cohort.
  logMAR
    number analyzed (Participants) | 183 | 175 | 0 | 0 | 358
    (all) | 0.05 (0.06) | 0.04 (0.05) |  |  | 0.04 (0.05)
Spectacle Wear [Count of Participants; unit: Participants] | 42 | 38 | 5 | 9 | 94
Preschool Randot Near Stereoacuity (arcsec) [Count of Participants; unit: Participants] — Stereoacuity scores (seconds of arc) were calculated based on the Randot Preschool stereoacuity test (scores: 800, 400, 200, 100, 60 and 40). Seconds of arc refers to the visual angle that is being measured in order to determine depth perception. Lower scores indicate better stereoacuity. Population: This measure was used exclusively with the older cohort, no data reported on this characteristic for the younger cohort.
  Participants
    40: number analyzed (Participants) | 183 | 175 | 0 | 0 | 358
    40 | 75 | 69 |  |  | 144
    60: number analyzed (Participants) | 183 | 175 | 0 | 0 | 358
    60 | 39 | 43 |  |  | 82
    100: number analyzed (Participants) | 183 | 175 | 0 | 0 | 358
    100 | 43 | 25 |  |  | 68
    200: number analyzed (Participants) | 183 | 175 | 0 | 0 | 358
    200 | 19 | 16 |  |  | 35
    400: number analyzed (Participants) | 183 | 175 | 0 | 0 | 358
    400 | 7 | 22 |  |  | 29
Preschool Randot Near Stereoacuity (arcsec) [Mean (Standard Deviation); unit: log arcsec] — Stereoacuity scores (seconds of arc, or arcsec) were calculated based on the Randot Preschool stereoacuity test (scores: 800, 400, 200, 100, 60 and 40). Seconds of arc refers to the visual angle that is being measured in order to determine depth perception. Lower scores indicate better stereoacuity.
  A logarithm base 10 transformation was used to convert stereoacuity scores to the log scale to calculate descriptive statistics (reported as log of seconds of arc, or log arcsec). Population: This measure was used exclusively with the older cohort, no data reported on this characteristic for the younger cohort.
  log arcsec
    number analyzed (Participants) | 183 | 175 | 0 | 0 | 358
    (all) | 1.84 (0.27) | 1.89 (0.34) |  |  | 1.87 (0.31)
Distance Randot Stereoacuity (arcsec) [Count of Participants; unit: Participants] — Stereoacuity scores (seconds of arc, or arcsec) were calculated based on the Randot Preschool stereoacuity test (scores: 800, 400, 200, 100, 60 and 40). Seconds of arc refers to the visual angle that is being measured in order to determine depth perception. Lower scores indicate better stereoacuity. Population: This measure was used exclusively with the older cohort, no data reported on this characteristic for the younger cohort.
  Participants
    60: number analyzed (Participants) | 183 | 175 | 0 | 0 | 358
    60 | 64 | 77 |  |  | 141
    100: number analyzed (Participants) | 183 | 175 | 0 | 0 | 358
    100 | 39 | 38 |  |  | 77
    200: number analyzed (Participants) | 183 | 175 | 0 | 0 | 358
    200 | 30 | 23 |  |  | 53
    400: number analyzed (Participants) | 183 | 175 | 0 | 0 | 358
    400 | 18 | 20 |  |  | 38
    Nil: number analyzed (Participants) | 183 | 175 | 0 | 0 | 358
    Nil | 28 | 16 |  |  | 44
Distance Randot Stereoacuity (arcsec) [Mean (Standard Deviation); unit: log arcsec] — Stereoacuity scores (seconds of arc, or arcsec) were calculated based on the Randot Preschool stereoacuity test (scores: 800, 400, 200, 100, 60 and 40). Seconds of arc refers to the visual angle that is being measured in order to determine depth perception. Lower scores indicate better stereoacuity.
  A logarithm base 10 transformation was used to convert stereoacuity scores to the log scale to calculate descriptive statistics (reported as log of seconds of arc, or log arcsec). Population: This measure was used exclusively with the older cohort, no data reported on this characteristic for the younger cohort.
  log arcsec
    number analyzed (Participants) | 183 | 175 | 0 | 0 | 358
    (all) | 2.22 (0.50) | 2.12 (0.44) |  |  | 2.17 (0.47)
Exotropia Type [Count of Participants; unit: Participants] — AC/A= accommodative convergence to accommodation ratio
  Participants
    Basic | 127 | 119 | 61 | 71 | 378
    Convergence insufﬁciency | 5 | 0 | 2 | 1 | 8
    High AC/A | 4 | 7 | 2 | 0 | 13
    Pseudodivergence excess | 39 | 39 | 26 | 24 | 128
    True divergence excess | 7 | 10 | 5 | 8 | 30
    Missing exotropia classification | 1 | 0 | 1 | 0 | 2
Deviation Type [Count of Participants; unit: Participants]
  Distance: Constant exotropia | 9 | 8 | 9 | 3 | 29
  Distance: Intermittent exotropia | 174 | 167 | 88 | 101 | 530
  Distance: Exophoria | 0 | 0 | 0 | 0 | 0
  Distance: No Exodeviation | 0 | 0 | 0 | 0 | 0
  Near: Constant exotropia | 1 | 1 | 0 | 0 | 2
  Near: Intermittent exotropia | 129 | 119 | 69 | 72 | 389
  Near: Exophoria | 49 | 44 | 21 | 21 | 135
  Near: No Exodeviation | 4 | 11 | 7 | 11 | 33
Exotropia (∆) by Simultaneous Prism Cover Test (SPCT) [Count of Participants; unit: Participants] — The Simultaneous Prism and Cover Test (SPCT) is performed by covering the fixating eye at the same time the prism is placed in front of the deviating eye. Prism diopters are the measure. Population: One participant was missing SPCT at near
  Participants
    Distance: 0 (no measureable tropia) | 48 | 50 | 28 | 41 | 167
    Distance: 1-9 | 15 | 18 | 8 | 7 | 48
    Distance: 10-14 | 18 | 12 | 4 | 5 | 39
    Distance: 16-18 | 30 | 29 | 8 | 13 | 80
    Distance: 20-25 | 57 | 47 | 30 | 21 | 155
    Distance: 30-35 | 13 | 15 | 16 | 12 | 56
    Distance: 40-50 | 2 | 4 | 3 | 3 | 12
    Distance: >50 | 0 | 0 | 0 | 2 | 2
    Near: number analyzed (Participants) | 183 | 175 | 97 | 103 | 558
    Near: 0 (no measureable tropia) | 108 | 108 | 63 | 75 | 354
    Near: 1-9 | 23 | 27 | 11 | 8 | 69
    Near: 10-14 | 21 | 11 | 4 | 3 | 39
    Near: 16-18 | 13 | 12 | 3 | 4 | 32
    Near: 20-25 | 14 | 9 | 12 | 9 | 44
    Near: 30-35 | 4 | 5 | 3 | 3 | 15
    Near: 40-50 | 0 | 3 | 1 | 1 | 5
    Near: >50 | 0 | 0 | 0 | 0 | 0
Average Exotropia (∆) by SPCT [Median (Full Range); unit: Prism Diopters] — The Simultaneous Prism and Cover Test (SPCT) is performed by covering the fixating eye at the same time the prism is placed in front of the deviating eye. Prism diopters are the measure.
  Prism Diopters
    Distance | 16 [0 to 45] | 16 [0 to 45] | 20 [0 to 50] | 14 [0 to 50] | 16 [0 to 50]
    Near | 0 [0 to 30] | 0 [0 to 45] | 0 [0 to 45] | 0 [0 to 40] | 0 [0 to 45]
Exodeviation (∆) by Prism and Alternate Cover Test (PACT) [Count of Participants; unit: Participants] — The prism and alternate cover test (PACT) is used to measure the angle of strabismus, or deviation, in prism diopters. This is measured separately at distance and at near. Smaller numbers are better because they indicate a smaller angle of deviation.
  Participants
    Distance: No exodeviation (orthophoria) | 0 | 0 | 0 | 0 | 0
    Distance: 1-9 | 0 | 0 | 00 | 0 | 0
    Distance: 10-14 | 7 | 11 | 0 | 0 | 18
    Distance: 16-18 | 34 | 33 | 9 | 14 | 90
    Distance: 20-25 | 101 | 87 | 44 | 44 | 276
    Distance: 30-35 | 35 | 39 | 39 | 36 | 149
    Distance: 40-45 | 5 | 5 | 3 | 8 | 21
    Distance: ≥50 | 1 | 0 | 2 | 2 | 5
    Near: No exodeviation (orthophoria) | 6 | 7 | 9 | 13 | 35
    Near: 1-9 | 19 | 31 | 7 | 8 | 65
    Near: 10-14 | 49 | 45 | 24 | 15 | 133
    Near: 16-18 | 32 | 24 | 9 | 13 | 78
    Near: 20-25 | 52 | 48 | 30 | 30 | 160
    Near: 30-35 | 21 | 15 | 14 | 18 | 68
    Near: 40-45 | 4 | 5 | 3 | 5 | 17
    Near: ≥50 | 0 | 0 | 1 | 2 | 3
Average Exodeviation (∆) by PACT [Mean (Standard Deviation); unit: Prism Diopters] — The prism and alternate cover test (PACT) is used to measure the angle of strabismus, or deviation, in prism diopters. This is measured separately at distance and at near. Smaller numbers are better because they indicate a smaller angle of deviation.
  Prism Diopters
    Distance | 23.3 (6.7) | 23.6 (6.7) | 27.4 (7.1) | 27.2 (8.2) | 24.8 (7.3)
    Near | 18.0 (8.9) | 16.7 (9.3) | 18.1 (10.8) | 19.4 (12.1) | 17.8 (10.0)
Exotropia control score [Count of Participants; unit: Participants] — Numeric values for exotropia control were assigned so that the following categories were created:
  Not applicable (no exodeviation) 0: No exotropia unless dissociated, recovers <1 secs (phoria)
  1. No exotropia unless dissociated, recovers 1-5 secs
  2. No exotropia unless dissociated, recovers >5 secs
  3. Exotropia <50% of 30-second observation
  4. Exotropia >50% of 30-second observation
  5. Constant exotropia
  Lower scores indicate better control.
  Participants
    Distance: No exodeviation | 0 | 0 | 0 | 0 | 0
    Distance: No XT unless dissociated, recovers <1 sec | 5 | 5 | 2 | 2 | 14
    Distance: No XT unless dissociated, recovers 1-5 sec | 34 | 47 | 18 | 27 | 126
    Distance: No XT unless dissociated, recovers >5 sec | 71 | 56 | 38 | 33 | 198
    Distance: XT <50% of 30-seconds | 40 | 37 | 19 | 27 | 123
    Distance: XT >50% of 30-seconds | 21 | 19 | 11 | 11 | 62
    Distance: Constant XT | 12 | 11 | 9 | 4 | 36
    Near: No exodeviation | 5 | 7 | 3 | 10 | 25
    Near: No XT unless dissociated, recovers <1 sec | 58 | 58 | 31 | 28 | 175
    Near: No XT unless dissociated, recovers 1-5 sec | 71 | 63 | 30 | 39 | 203
    Near: No XT unless dissociated, recovers >5 sec | 28 | 26 | 17 | 15 | 86
    Near: XT <50% of 30-seconds | 18 | 14 | 12 | 11 | 55
    Near: XT >50% of 30-seconds | 2 | 7 | 4 | 1 | 14
    Near: Constant XT | 1 | 0 | 0 | 0 | 1
Average Exotropia Control Score [Mean (Standard Deviation); unit: scores on a scale] — Numeric values for exotropia control were assigned so that the following categories were created:
  Not applicable (no exodeviation) 0: No exotropia unless dissociated, recovers <1 secs (phoria)
  1. No exotropia unless dissociated, recovers 1-5 secs
  2. No exotropia unless dissociated, recovers >5 secs
  3. Exotropia <50% of 30-second observation
  4. Exotropia >50% of 30-second observation
  5. Constant exotropia
  Lower scores indicate better control.
  scores on a scale
    Distance | 2.4 (1.2) | 2.3 (1.2) | 2.5 (1.2) | 2.3 (1.1) | 2.4 (1.2)
    Near | 1.1 (1.0) | 1.1 (1.1) | 1.2 (1.2) | 1.0 (1.0) | 1.1 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Deterioration by 6 Months - Older Cohort
Description: The primary outcome measure for this study was whether the participant's condition had deteriorated within 6 months after randomization. Deterioration was defined as meeting one or both of the following criteria during a masked examination at either the 3-month or 6-month visit: 1) a constant exotropia (throughout the exam) of 10∆ or greater at distance and near by SPCT, confirmed by a retest, or 2) loss of near stereoacuity of 2 octaves (0.6 log arcsec) or more from the better of a test and retest of Preschool Randot stereoacuity at baseline, confirmed by a retest. In addition, participants were classified as deteriorated for the primary analysis if they started using non-randomized treatment (i.e., any treatment in the observation group; any treatment other than patching in the patching group) without first meeting one of the two protocol-specified deterioration criteria.
Time Frame: 6 months
Population: Previously untreated children aged 3 to <11 years. The 6-month primary outcome visit was completed by 165 participants (90%) in the observation group, and by 159 participants (91%) in the patching group.
Measure: Count of Participants; unit: Participants
Groups:
- Older Cohort Observation Group: Older cohort patients randomized to the observation group will receive no treatment (other than refractive correction).
- Older Cohort Occlusion Therapy Group: Occlusion treatment: older cohort patients randomized to the occlusion treatment group will receive occlusion (patching) for 3 hours per day for at least 3 months. Choice of which eye to occlude, or whether to alternate daily, is at investigator's discretion.
Arm/Group | Older Cohort Observation Group | Older Cohort Occlusion Therapy Group
Number analyzed (Participants) | 165 | 159
Participants
  Formal deterioration criteria met | 10 | 1
  Constant exotropia >= 10 PD at distance and near | 7 | 1
  Stereoacuity worsening of >= 2 octaves | 1 | 0
  Both criteria | 0 | 0
  Started treatment w/o meeting criteria | 3 | 0
Statistical Analysis 1: Comparison: Older Cohort Observation Group vs Older Cohort Occlusion Therapy Group; Test type: Superiority; p = 0.004, One-sided Barnard's Test; Risk Difference (RD) = 0.054, 95% CI 1-sided [lower limit 0.020]

2. Primary Outcome: Deterioration by 3 Years - Older Cohort
Description: The primary outcome measure for this study was whether the participant's condition had deteriorated within 3 years after randomization. Deterioration was defined as meeting one or both of the following criteria during any masked examination between 3 months and 3 years after randomization: 1) a constant exotropia (throughout the exam) of 10∆ or greater at distance and near by SPCT, confirmed by a retest, or 2) loss of near stereoacuity of 2 octaves (0.6 log arcsec) or more from the better of a test and retest of Preschool Randot stereoacuity at baseline, confirmed by a retest. In addition, participants were classified as deteriorated for the primary analysis if they started using non-randomized treatment (i.e., any treatment in the observation group; any treatment other than patching in the patching group) without first meeting one of the two protocol-specified deterioration criteria.
Time Frame: 3 years
Population: The clinical trial ended after 6 months, after which the purpose of the study was to observe the natural history of patients in the Observation arm. Because only half the occlusion group underwent further occlusion between 6 months and 3 years, the long-term occlusion group data was not felt to be of value, and there are no plans for its analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Older Cohort Occlusion Therapy Group: This group was not reported on. The clinical trial ended after 6 months, after which the purpose of the study was to observe the natural history of patients in the Observation arm. No data were collected from participants from 6 months to 3 years, and there are no plans for analysis.
Arm/Group | Older Cohort Observation Group | Older Cohort Occlusion Therapy Group
Number analyzed (Participants) | 183 | 0
Participants | 25 | 0
Statistical Analysis 1: Comparison: Older Cohort Observation Group; Test type: Other; cumulative probability = .15, 95% CI 2-sided [.10 to .22] — Kaplan-Meier estimate of cumulative probability of deterioration by 3 years

3. Primary Outcome: Deterioration by 6 Months - Younger Cohort
Description: The primary outcome measure was deterioration of the intermittent exotropia (IXT) within 6 months after randomization. Motor deterioration was deﬁned as a constant exotropia of 10 D or more at distance and near by SPCT, conﬁrmed by a retest, at either the 3- or 6-month visit.
Time Frame: 6 months
Population: Previously untreated children aged 12 to 35 months. Motor deterioration was measured by simultaneous prism and cover test.
Measure: Count of Participants; unit: Participants
Arm/Group | Younger Cohort Observation Group | Younger Cohort Occlusion Therapy Group
Number analyzed (Participants) | 87 | 90
Participants
  Deterioration | 4 | 2
  Constant exotropia >= 10 PD at distance and near | 2 | 2
  Started nonprotocol tmt w/o motor deterioration | 2 | 0
Statistical Analysis 1: Comparison: Younger Cohort Observation Group vs Younger Cohort Occlusion Therapy Group; Test type: Superiority; p = 0.27, One-sided Barnard's Test; Risk Difference (RD) = 0.024, 95% CI 2-sided [-0.038 to 0.094]

4. Primary Outcome: Deterioration by 3 Years - Younger Cohort
Description: The primary outcome measure was deterioration of the intermittent exotropia (IXT) within 6 months after randomization. Motor deterioration was deﬁned as a constant exotropia of 10 D or more at distance and near by SPCT, conﬁrmed by a retest, during any masked examination between 3 months and 3 years after randomization.
Time Frame: 3 years
Population: The younger cohort occlusion therapy group was not reported on. The clinical trial ended after 6 months, after which the purpose of the study was to observe the natural history of patients in the Observation arm. No data were collected from participants from 6 months to 3 years, and there are no plans for analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Younger Cohort Occlusion Therapy Group: This group was not reported on. The clinical trial ended after 6 months, after which the purpose of the study was to observe the natural history of patients in the Observation arm. No data were collected from participants from 6 months to 3 years, and there are no plans for analysis.
Arm/Group | Younger Cohort Observation Group | Younger Cohort Occlusion Therapy Group
Number analyzed (Participants) | 97 | 0
Participants | 24 | 0

5. Secondary Outcome: Distance Stereoacuity - 3 Years
Description: Stereoacuity scores (seconds of arc) were calculated based on the Randot Preschool stereoacuity test (scores: 800, 400, 200, 100, 60 and 40). Seconds of arc refers to the visual angle that is being measured in order to determine depth perception. Lower scores indicate better stereoacuity.
  A logarithm base 10 transformation was used to convert stereoacuity scores to the log scale to calculate descriptive statistics (reported as log of seconds of arc, or log arcsec). The stereoacuity at distance is reported at 3 years, as is the change in distance stereoacuity from baseline to 3 years. Both were reported as log of seconds of arc, or log arcsec. For change in stereo, positive change indicates improvement in stereo.
Time Frame: Between baseline and 3 years
Population: Since only half the occlusion group underwent further occlusion between 6 months and 3 years, the long-term occlusion group data was not felt to be of value, and there are no plans for its analysis. For the observation group, the number reported is those who completed the 3-Year visit and had not been prescribed treatment anytime during the study.
Measure: Mean (Standard Deviation); unit: log arsec
Groups:
- Older Cohort Occlusion Group: This group was not reported on. The clinical trial ended after 6 months, after which the purpose of the study was to observe the natural history of patients in the Observation arm. No data were collected from participants from 6 months to 3 years, and there are no plans for analysis.
Arm/Group | Older Cohort Observation Group | Older Cohort Occlusion Group
Number analyzed (Participants) | 132 | 0
log arsec
  At 3 Years | 2.03 (0.36) |
  Change between baseline and 3 years | 0.14 (0.40) |
Statistical Analysis 1: Comparison: Older Cohort Observation Group; P-value for the change between baseline and 3 years. Two-sided p values for comparisons of continuous outcomes are from analysis of covariance models adjusting for the baseline level of the outcome; Test type: Other; p < .001, ANCOVA

6. Secondary Outcome: Near Stereoacuity - 6 Months
Description: Stereoacuity scores (seconds of arc) were calculated based on the Randot Preschool stereoacuity test (scores: 800, 400, 200, 100, 60 and 40). Seconds of arc refers to the visual angle that is being measured in order to determine depth perception. Lower scores indicate better stereoacuity.
  A logarithm base 10 transformation was used to convert stereoacuity scores to the log scale to calculate descriptive statistics (reported as log of seconds of arc, or log arcsec). The stereoacuity at near is reported at 3 years, as is the change in near stereoacuity from baseline to 3 years. Both were reported as log of seconds of arc, or log arcsec.
  Outcome based on initial testing regardless of whether a retest was completed for suspected deterioration. Change is calculated as baseline level minus 6-month level. For change in stereo, positive change indicates improvement in stereo.
Time Frame: 6 months
Population: Stereoacuity data is missing for 2 observation group participants because it was not tested at the visit at which treatment was started in the absence of meeting deterioration criteria. The 6-month primary outcome visit was completed by 165 participants (90%) in the observation group, and by 159 participants (91%) in the patching group.
Measure: Mean (Standard Deviation); unit: log arsec
Arm/Group | Older Cohort Observation Group | Older Cohort Occlusion Therapy Group
Number analyzed (Participants) | 165 | 159
log arsec
  At 6 months | 1.84 (0.33) | 1.84 (0.31)
  Change between Baseline and 6 months | 0.00 (0.32) | 0.06 (0.30)
Statistical Analysis 1: Comparison: Older Cohort Observation Group vs Older Cohort Occlusion Therapy Group; Two-sided p values for comparisons of continuous outcomes are from analysis of covariance models adjusting for the baseline level of the outcome; P values for comparisons of binary outcomes are from logistic regression models adjusting for the baseline level of the outcome; Test type: Other; p = 0.38, ANCOVA

7. Secondary Outcome: Near Stereoacuity - 3 Years
Description: Stereoacuity scores (seconds of arc) were calculated based on the Randot Preschool stereoacuity test (scores: 800, 400, 200, 100, 60 and 40). Seconds of arc refers to the visual angle that is being measured in order to determine depth perception. Lower scores indicate better stereoacuity.
  A logarithm base 10 transformation was used to convert stereoacuity scores to the log scale to calculate descriptive statistics (reported as log of seconds of arc, or log arcsec). The stereoacuity at near is reported at 3 years, as is the change in near stereoacuity from baseline to 3 years. Both were reported as log of seconds of arc, or log arcsec. For change in stereo, positive change indicates improvement in stereo.
Time Frame: between baseline and 3 years
Population: The older cohort occlusion therapy group was not reported on. The clinical trial ended after 6 months, after which the purpose of the study was to observe the natural history of patients in the Observation arm. No data were collected from participants from 6 months to 3 years, and there are no plans for analysis.
Measure: Mean (Standard Deviation); unit: log arcsec
Arm/Group | Older Cohort Observation Group | Older Cohort Occlusion Therapy Group
Number analyzed (Participants) | 132 | 0
log arcsec
  At 3 Years | 1.7 (0.21) |
  Change between Baseline and 3 Years | 0.14 (0.29) |
Statistical Analysis 1: Comparison: Older Cohort Observation Group; [analysis description as in outcome 5, analysis 1]; Test type: Other; p < .001, ANCOVA

8. Secondary Outcome: Exotropia Control at Distance - 6 Months
Description: Change in control is calculated as baseline level minus 3-year level, so positive change = improvement. Scale Range: 0 to 5. Improvement in control was defined as an improvement of 3 points based on the 3-point threshold for real change.
  Numeric values for exotropia control were assigned so that the following categories were created:
  Not applicable (no exodeviation) 0: No exotropia unless dissociated, recovers <1 secs (phoria)
  1. No exotropia unless dissociated, recovers 1-5 secs
  2. No exotropia unless dissociated, recovers >5 secs
  3. Exotropia <50% of 30-second observation
  4. Exotropia >50% of 30-second observation
  5. Constant exotropia
  Lower scores indicate better control.
Time Frame: 6 months
Population: For the Older Cohort, the 6-month primary outcome visit was completed by 165 participants (90%) in the observation group, and by 159 participants (91%) in the patching group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Older Cohort Observation Group | Older Cohort Occlusion Therapy Group | Younger Cohort Observation Group | Younger Cohort Occlusion Therapy Group
Number analyzed (Participants) | 165 | 159 | 87 | 90
score on a scale
  At 6 months | 2.3 (1.4) | 2.0 (1.2) | 2.8 (1.3) | 2.3 (1.5)
  Change between Baseline and 6 months | 0.1 (1.4) | 0.3 (1.4) | -0.3 (1.3) | 0.1 (1.5)
Statistical Analysis 1: Comparison: Older Cohort Observation Group vs Older Cohort Occlusion Therapy Group; P-value for the change between baseline and 6 months in the Older cohort. Two-sided p values for comparisons of continuous outcomes are from analysis of covariance models adjusting for the baseline level of the outcome; Test type: Other; p = 0.09, ANCOVA
Statistical Analysis 2: Comparison: Younger Cohort Observation Group vs Younger Cohort Occlusion Therapy Group; P-value for the change between baseline and 6 months in the Younger cohort. Two-sided p values for comparisons of continuous outcomes are from analysis of covariance models adjusting for the baseline level of the outcome; Test type: Other; p = 0.02, ANCOVA

9. Secondary Outcome: Exotropia Control at Distance - 3 Years
Description: as for outcome 8
Time Frame: 3 years
Population: Since only half the occlusion group underwent further occlusion between 6 months and 3 years, the long-term occlusion group data was not felt to be of value, and there are no plans for its analysis. For the observation groups, the number reported is those who completed the 3-Year visit and had not been prescribed treatment anytime during the study.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Younger Cohort Occlusion Group: This group was not reported on. The clinical trial ended after 6 months, after which the purpose of the study was to observe the natural history of patients in the Observation arm. No data were collected from participants from 6 months to 3 years, and there are no plans for analysis.
Arm/Group | Older Cohort Observation Group | Older Cohort Occlusion Group | Younger Cohort Observation Group | Younger Cohort Occlusion Group
Number analyzed (Participants) | 132 | 0 | 53 | 0
score on a scale
  At 3 Years | 1.8 (1.4) |  | 2.2 (1.5) |
  Change between Baseline and 3 Years | 0.6 (1.5) |  | 0.2 (1.4) |
Statistical Analysis 1: Comparison: Older Cohort Observation Group; P-value for the change between baseline and 3 Years in the Older cohort. Two-sided p values for comparisons of continuous outcomes are from analysis of covariance models adjusting for the baseline level of the outcome; Test type: Other; p < .001, ANCOVA
Statistical Analysis 2: Comparison: Younger Cohort Observation Group; P-value for the change between baseline and 3 Years in the Younger cohort. Two-sided p values for comparisons of continuous outcomes are from analysis of covariance models adjusting for the baseline level of the outcome; Test type: Other; p = 0.33, ANCOVA

10. Secondary Outcome: Exotropia Control at Near - 6 Months
Description: as for outcome 8
Time Frame: 6 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Older Cohort Observation Group | Older Cohort Occlusion Therapy Group | Younger Cohort Observation Group | Younger Cohort Occlusion Therapy Group
Number analyzed (Participants) | 165 | 159 | 87 | 90
score on a scale
  A 6 months | 1.2 (1.1) | 0.9 (1.1) | 1.4 (1.4) | 1.1 (1.4)
  Change between Baseline and 6 months | -0.2 (1.1) | 0.1 (1.1) | -0.3 (1.1) | -0.1 (1.3)
Statistical Analysis 1: Comparison: Older Cohort Observation Group vs Older Cohort Occlusion Therapy Group; [analysis description as in outcome 8, analysis 1]; Test type: Other; p = 0.013, ANCOVA
Statistical Analysis 2: Comparison: Younger Cohort Observation Group vs Younger Cohort Occlusion Therapy Group; [analysis description as in outcome 8, analysis 2]; Test type: Other; p = 0.26, ANCOVA

11. Secondary Outcome: Exotropia Control at Near - 3 Years
Description: as for outcome 8
Time Frame: 3 years
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Older Cohort Observation Group | Older Cohort Occlusion Group | Younger Cohort Observation Group | Younger Cohort Occlusion Group
Number analyzed (Participants) | 132 | 0 | 53 | 0
score on a scale
  At 3 Years | 0.9 (1.1) |  | 1.0 (1.4) |
  Change between Baseline and 3 Years | 0.1 (1.2) |  | 0.1 (1.4) |
Statistical Analysis 1: Comparison: Older Cohort Observation Group; [analysis description as in outcome 9, analysis 1]; Test type: Other; p = 0.42, ANCOVA
Statistical Analysis 2: Comparison: Younger Cohort Observation Group; [analysis description as in outcome 9, analysis 2]; Test type: Other; p = 0.61, ANCOVA

12. Secondary Outcome: PACT Exodeviation at Distance - 6 Months
Description: The prism and alternate cover test (PACT) is used to measure the angle of strabismus, or deviation, in prism diopters. This is measured separately at distance and at near. Smaller numbers are better because they indicate a smaller angle of deviation. For change in PACT, positive change indicates improvement (i.e. decrease in angle over time).
  log arcsec = logarithm of seconds of arc; Δ = prism diopter
Time Frame: 6 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: prism diopters
Arm/Group | Older Cohort Observation Group | Older Cohort Occlusion Therapy Group | Younger Cohort Observation Group | Younger Cohort Occlusion Therapy Group
Number analyzed (Participants) | 165 | 159 | 87 | 90
prism diopters
  At 6 months | 23.8 (7.8) | 22.2 (7.4) | 27.9 (8.2) | 24.9 (9.4)
  Change between Baseline and 6 months | -0.3 (6.8) | 1.4 (5.8) | -0.6 (8.1) | 2.0 (8.6)
Statistical Analysis 1: Comparison: Older Cohort Observation Group vs Older Cohort Occlusion Therapy Group; [analysis description as in outcome 8, analysis 1]; Test type: Other; p = 0.012, ANCOVA
Statistical Analysis 2: Comparison: Younger Cohort Observation Group vs Younger Cohort Occlusion Therapy Group; [analysis description as in outcome 8, analysis 2]; Test type: Other; p = 0.02, ANCOVA

13. Secondary Outcome: PACT at Distance - 3 Years
Description: The prism and alternate cover test (PACT) is used to measure the angle of strabismus, or deviation, in prism diopters. This is measured separately at distance and at near. Smaller numbers are better because they indicate a smaller angle of deviation. For change in PACT, positive change indicates improvement (i.e. decrease in angle over time). Improvement in PACT at distance was defined as a decrease of ≥8∆ because this amount exceed the repeatability coefficient of 7.2∆ for PACT angles larger than 20∆ at distance.
  log arcsec = logarithm of seconds of arc; Δ = prism diopter
Time Frame: 3 years
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: prism diopters
Arm/Group | Older Cohort Observation Group | Older Cohort Occlusion Group | Younger Cohort Observation Group | Younger Cohort Occlusion Group
Number analyzed (Participants) | 132 | 0 | 53 | 0
prism diopters
  At 3 Years | 21.0 (8.7) |  | 23.4 (9.5) |
  Change between Baseline and 3 Years | 2.2 (8.3) |  | 3.6 (10.4) |
Statistical Analysis 1: Comparison: Older Cohort Observation Group; [analysis description as in outcome 9, analysis 1]; Test type: Other; p = .002, ANCOVA
Statistical Analysis 2: Comparison: Younger Cohort Observation Group; [analysis description as in outcome 9, analysis 2]; Test type: Other; p = 0.01, ANCOVA

14. Secondary Outcome: PACT at Near - 6 Months
Description: as for outcome 12
Time Frame: 6 months
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: prism diopters
Arm/Group | Older Cohort Observation Group | Older Cohort Occlusion Therapy Group | Younger Cohort Observation Group | Younger Cohort Occlusion Therapy Group
Number analyzed (Participants) | 165 | 159 | 87 | 90
prism diopters
  At 6 months | 17.6 (9.6) | 15.4 (10.1) | 19.3 (9.6) | 17.0 (12.2)
  Change between Baseline and 6 months | 0.5 (7.8) | 1.5 (8.0) | -1.8 (11.4) | 0.9 (12.8)
Statistical Analysis 1: Comparison: Older Cohort Observation Group vs Older Cohort Occlusion Therapy Group; [analysis description as in outcome 8, analysis 1]; Test type: Other; p = 0.11, ANCOVA
Statistical Analysis 2: Comparison: Younger Cohort Observation Group vs Younger Cohort Occlusion Therapy Group; [analysis description as in outcome 8, analysis 2]; Test type: Other; p = 0.10, ANCOVA

15. Secondary Outcome: PACT at Near - 3 Years
Description: The prism and alternate cover test (PACT) is used to measure the angle of strabismus, or deviation, in prism diopters. This is measured separately at distance and at near. Smaller numbers are better because they indicate a smaller angle of deviation. For change in PACT, positive change indicates improvement (i.e. decrease in angle over time).
  Improvement in PACT at near was defined as a decrease of ≥13∆ because this amount exceed the repeatability coefficient of 12.8∆ for PACT angles larger than 20∆ at near.
  log arcsec = logarithm of seconds of arc; Δ = prism diopter
Time Frame: 3 years
Population: as for outcome 9
Measure: Mean (Standard Deviation); unit: prism diopters
Arm/Group | Older Cohort Observation Group | Older Cohort Occlusion Group | Younger Cohort Observation Group | Younger Cohort Occlusion Group
Number analyzed (Participants) | 132 | 0 | 53 | 0
prism diopters
  At 3 Years | 17.0 (10.1) |  | 14.9 (10.3) |
  Change between Baseline and 3 Years | 0.4 (9.3) |  | 2.8 (12.0) |
Statistical Analysis 1: Comparison: Older Cohort Observation Group; [analysis description as in outcome 9, analysis 1]; Test type: Other; p = 0.60, ANCOVA
Statistical Analysis 2: Comparison: Younger Cohort Observation Group; [analysis description as in outcome 9, analysis 2]; Test type: Other; p = 0.09, ANCOVA

ADVERSE EVENTS:
Arm/Group | Older Cohort Observation Group | Older Cohort Occlusion Therapy Group | Younger Cohort Observation Group | Younger Cohort Occlusion Therapy Group
All-Cause Mortality (participants affected / at risk) | 0/183 | 0/175 | 0/97 | 0/104
Serious Adverse Events (participants affected / at risk) | 0/183 | 0/175 | 0/97 | 0/104
Other Adverse Events (participants affected / at risk) | 0/183 | 0/175 | 0/97 | 0/104

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No